CLINICAL TRIAL: NCT06940531
Title: Identifying the Causes and Risk Factors of Pulmonary Exacerbations in Cystic Fibrosis
Acronym: CF-Tracker
Status: Not yet recruiting | Type: Observational
Sponsor: Alexander Horsley (Other)
Responsible Party: Sponsor-Investigator, Alexander Horsley, Professor of Respiratory Medicine and Honorary Consultant, University of Manchester
Organization: University of Manchester (Other)
Other Study IDs: 338539
Record Dates: First submitted 2025-04-01; First posted 2025-04-23 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Cystic Fibrosis (CF); Cystic Fibrosis Pulmonary Exacerbation
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Spirometry
  * Impulse oscillometry
  * Venous blood draw
  * Saliva sample
  * Sputum sample
  * Cough swab
  * Urine Sample
  * Nose and throat swab
  * Exhaled volatiles (VOCs)
  * Exhaled nitric oxide (FeNO)
  * Nasal liquid sample
  * Rectal swabs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Group A: 200 adults with CF (16 years or older) will be recruited to Group A. Group A participants will have a single in-person visit, at the start of the study. Clinical data, including lung function (spirometry), venous blood draw, sweat chloride, saliva sample and finger-prick dried blood spot sample, sputum, nasal liquid sample and urine sample and demographic data will be collected. The study will run for 12 months. Home sampling kit, consisting of 13 home sampling boxes and 3 additional exacerbation boxes, will be provided for participants to collect in-home sampling for the first 6 months fortnightly. The 3 additional exacerbation boxes will be provided for posting additional set of samples when unwell. There will be questionnaires to complete to remotely monitor the adherence to the protocol. The study app will be set up to provide reminders and aid study adherence and timely return of samples.
- Group B: 100 adults with CF (16 years or older) will be recruited to Group B. Group B will only be offered at 5 specialist CF centres (Manchester, Cardiff, Newcastle, Leeds, Liverpool). This follows the same format as Group A but includes additional face to face visits at 1 and 6 months, and the invitation to return for additional samples if unwell. In Group B, those attending the Manchester clinic will have the option of taking part in a 12 month home environmental and pollution monitoring and sleep monitoring (both optional arms).
- Paediatric Pilot Study: An additional feasibility cohort of up to 25 paediatric patients (aged 5-15 years) will be included. This will open in up to 4 centres who are already running the adult study. The basic study protocol will be the same as for Group A, with a single patient visit at the start of the study and the remainder of the assessments from home monitoring. Parental consent, participant consent and assent will be obtained.
- Healthy Volunteers: 40 healthy volunteers will be recruited to ensure that the investigators have reference values for some of the established and experimental biomarkers. Clinical samples, including sputum, venous blood draw, nose and throat swabs, FeNo, VOCs and nasal liquid, and demographic information will be collected on a single occasion. Visits will take place at CRFs and are planned for the Manchester site only.

SUMMARY:
The CF-Tracker study is a community surveillance study, designed to understand the causes of exacerbations in people with cystic fibrosis (CF) (pwCF). These are episodes when pwCF become more unwell, typically characterised by increased cough, sputum, and breathlessness, and requiring prolonged courses of oral or intravenous antibiotics.

This observational study applies a two-tiered approach over 12 months. It will recruit 200 pwCF to Group A, and an additional 100 pwCF to Group B, which follows the same format but includes additional in-clinic sampling.

Participants will provide longitudinal clinical data and biological samples. Group B will be offered at 5 specialist CF centres (Manchester, Cardiff, Newcastle, Leeds, Liverpool), will include additional sampling methods at clinic visits, and additional scheduled clinic visits at 1 month and 6 months. Group B participants will be offered an in-person visit if they become unwell, so that samples can be collected before they start antibiotics. In Group B, those attending the Manchester clinic will have the option of taking part in a 12 month home environmental and pollution monitoring, and sleep monitoring (both optional arms).

A pilot study will test the practicalities of running the same protocol in a paediatric population. This will consist of up to 25 children with CF (5-15 years) attending a paediatric clinic in one of the four core centres. Up to 40 healthy volunteers will be recruited to provide samples on a single occasion as controls.

This study is funded by the Cystic Fibrosis Trust. This study is part of a wider programme of research, led by the PULSE-CF Innovation Hub (and hosted by the University of Manchester, www.pulse-cf.com). The aim of the Hub is that the data from CF-Tracker will support the delivery of a platform clinical trial to test exacerbation-prevention interventions in CF.

DETAILED DESCRIPTION:
Participants will be recruited by staff within the care of UK CF centres. Initial discussions will occur either during routine outpatient reviews, telephone consultations or during admissions. Consent will take place prior to any other procedures.

There will be four separate cohorts of participant

1. Group A participants will be 200 adults with CF (16 years or older) attending a UK adult CF centre taking part in the study
2. Group B participants will be 100 additional adults with CF attending one of the five core CF adult centres: Manchester, Leeds, Newcastle, Cardiff, Liverpool.
3. There will be a pilot study to test the practicalities of running the same protocol in a paediatric population. This will consist of up to 25 children with CF (5-16 years) attending a paediatric clinic in one of the five core centres.
4. In addition, the investigators will recruit up to 40 healthy volunteers to provide samples on a single occasion as controls.

Group A participants will have a single in-person visit, at the start of the study. Clinical data, including lung function (spirometry), venous blood draw, sweat chloride, saliva sample and finger-prick dried blood spot sample, sputum, nasal liquid sample and urine sample and demographic data will be collected. The study will run for 12 months. Home sampling kit, consisting of 13 home sampling boxes and 3 additional exacerbation boxes, will be provided for participants to collect in-home sampling for the first 6 months fortnightly. The 3 additional exacerbation boxes will be provided for posting additional set of samples when unwell. There will be questionnaires to complete to remotely monitor the adherence to the protocol. Study app ("Watson") will be set up to provide reminders and aid study adherence and timely return of samples.

Group B will only be offered at 5 specialist CF centres (Manchester, Cardiff, Newcastle, Leeds, Liverpool). This follows the same format as Group A but includes additional face to face visits at 1 and 6 months, and the invitation to return for additional samples if unwell. In Group B, those attending the Manchester clinic will have the option of taking part in a 12 month home environmental and pollution monitoring and sleep monitoring (both optional arms).

The investigators will include an additional feasibility cohort of up to 25 paediatric patients (aged 5-15 years). This will open in up to 4 centres who are already running the adult study. The basic study protocol will be the same as for Group A, with a single patient visit at the start of the study and the remainder of the assessments from home monitoring. Parental consent, participant consent and assent will be obtained.

In order to ensure that the investigators have reference values for some of the established and experimental biomarkers, the investigators will also collect samples from 40 healthy volunteers on a single occasion. Visits will take place at CRFs and are planned for the Manchester site only. Clinical samples, including sputum, venous blood draw, nose and throat swabs, FeNo, VOCs and nasal liquid, and demographic information will be collected.

ELIGIBILITY:
Inclusion Criteria:

For Adult Participants

1. Confirmed diagnosis of cystic fibrosis (CF), defined as presence of two pathogenic CF-causing CFTR mutations AND clinical features consistent with a diagnosis of CF, OR presence of at least one pathogenic CF-causing CFTR mutation AND sweat chloride (before use of CFTR modulators) >60mmol/L AND clinical features consistent with a diagnosis of CF.
2. Age ≥ 16 years and receiving care from a UK Adult Cystic Fibrosis Centre for main study. 5-16yrs for Paediatric pilot study (see below).
3. Have had at least 1 previous exacerbation of CF lung disease, treated with oral or intravenous antibiotics, in the previous 12 months.
4. Able to understand the patient information sheet, willing to consent to study protocol and to returning home samples
5. Has a home spirometry device and able to use this

   For those taking part in Group-B, additional inclusion criteria include
6. Willing to attend for additional face to face visits at 4 weeks, 26 weeks, and if they become unwell

   For those taking part in home monitoring (as part of Group-B at Manchester)
7. Has wireless internet at home
8. Willing to allow to home access to set up monitoring devices, collect these back in at end of study, and to carry out other visits to perform calibration or intermittent home air sampling.

For Paediatric Participants

1. Confirmed diagnosis of cystic fibrosis (CF), defined as presence of two pathogenic CF-causing CFTR mutations AND clinical features consistent with a diagnosis of CF, OR presence of at least one pathogenic CF-causing CFTR mutation AND sweat chloride (before use of CFTR modulators) >60mmol/L AND clinical features consistent with a diagnosis of CF.
2. Receiving care from an eligible Paediatric CF Centre.
3. Age 5-16 years
4. Have had at least 1 previous exacerbation of CF lung disease, treated with antibiotics.
5. Able to understand the study and/or willing to assent to study protocol.
6. Parents or guardians able to understand the study and willing to consent to take part, including helping with home sampling
7. Has a home spirometry device and able to use this

For Healthy Volunteers

1. Healthy subject, male or female, aged 16-65 years
2. No active lung condition, chronic inflammatory disorder or infection
3. Not been on antibiotics or anti-inflammatory agents of any sort (including inhaled or systemic corticosteroids) for at least 90 days.
4. No recent (defined as within the previous 4 weeks) acute viral symptoms
5. Willing to sign the consent form and provide the samples.

Exclusion Criteria:

1. Unable to produce sputum, spontaneous or induced, at visit 1. If subject is normally able to produce sputum and still wishes to take part, visit 1 can be repeated on up to two additional occasions if this is needed to obtain sputum sample.
2. For the first visit, participants should be clinically stable at the time of the visit. This is defined as no acute change in their baseline symptoms or presence of new viral symptoms. They should not be on additional antibiotics or anti-viral therapies for any reason (above their usual medications), and should have completed any such additional therapies at least 4 weeks prior to visit 1.
3. Subjects with infection with Mycobacteria tuberculosis
4. Subjects with active ABPA, defined as receiving treatment for ABPA currently or within the last 12 months, or those considered at risk of requiring treatment for ABPA in the next 12 months.
5. Subjects receiving long term oral steroids at an equivalent dose of 10mg or more per day of prednisolone.
6. Subjects receiving any other form of long term immune-suppressant therapy.
7. Subjects with non-tuberculous mycobacteria (NTM) infection who are undergoing active eradication therapy. Subjects with chronic NTM infection who are not on eradication therapy, and not expecting to start this within the next 12 months, are not excluded.
8. Subjects who are unable to complete home spirometry who have previously been shown poor adherence to home monitoring requests
9. Any other condition, co-morbidity or other feature that, in the opinion of the investigator would render the subject unable to complete the protocol or unsuitable for inclusion.
10. For home monitoring, any subject where the investigator or their team has concern about staff safety when performing home visits.

Patients taking part in other long term trials or observational studies are eligible to take part in CF-Tracker. Local investigators should judge whether the burden of additional research visits will be manageable.

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: United Kingdom
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-04-15 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Time to first exacerbation | 12 months
  Time (in days) to first exacerbation treated with oral or intravenous antibiotics is the primary outcome against which inflammatory marker data will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Manchester Adult Cystic Fibrosis Centre, Manchester University Hospitals NHS Foundation Trust, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Once collected and full anonymised, data will be made open to share based on FAIR data principles. Access to emerging datasets, or parts of datasets, is also possible based on a Data Access Application to the study team, which will be reviewed by the steering commitee.
Supporting Information: Study Protocol, Analytic Code
Time Frame: Details to be decided, but plan would be to make complete datasets open access.
Access Criteria: Data access is by application to the Steering Committee. For details on how to apply please email the study coordinator or PI

REFERENCES:
- See also: Hub website, with study pages — https://www.pulse-cf.com